CLINICAL TRIAL: NCT07145957
Title: Does Undergoing a Prehabilitation Protocol Aimed at Optimizing Scapulothoracic Mobility and Strengthening Improve Internal Rotation After Reverse Shoulder Arthroplasty? A Randomized Controlled Trial
Brief Title: Does Undergoing a Prehabilitation Protocol Aimed at Optimizing Scapulothoracic Mobility and Strengthening Improve Internal Rotation After Reverse Shoulder Arthroplasty?
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Shoulder and Elbow Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202501188
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Primary Reverse Total Shoulder Arthroplasty
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treatment (IRTx): IRTx group to complete the preoperative rehabilitation program
  Interventions: Other: Prehabilitation
- control (COS)

INTERVENTIONS:
Other: Prehabilitation — subjects randomized to the IRTx cohort will also be instructed by a Physical or Occupational Therapist to perform the exercises described in the RSA IR Prehab Exercise Protocol handout, 5-7 times per week for 6 weeks.
  Groups: treatment (IRTx)

SUMMARY:
Difficulty with internal rotation (IR) after reverse shoulder arthroplasty (RSA) is common. Current rehabilitation protocols may not optimize IR. The investigator's objective is to assess the impact of prehabilitation focused on IR strengthening and mobility on RSA outcomes. The investigators will perform a prospective, randomized control trial to achieve the specific aim: assessing range of motion, strength, patient-reported outcomes, and activities of daily living requiring internal rotation between control and prehabilitation cohorts, with the prehabilitation patients receiving 6 weeks of treatment.

DETAILED DESCRIPTION:
Reverse total shoulder arthroplasty (RSA) provides excellent restoration of overhead motion and pain relief, with durability demonstrated up to 20-years postoperatively.6 However, despite advancements in surgical technique and implants, internal rotation (IR) remains challenging for many patients after RSA, with a recent study demonstrating as many as 63% of patients reporting significant difficulty or inability to perform some activities of daily living (ADLs) requiring IR.5

Many studies have been conducted to identify demographic, surgical, and implant-related predictors of improved IR after RSA. To date, the only consistent predictor of superior IR after RSA in the literature is more favorable preoperative IR. Nearly all interventions that have been evaluated to improve IR after RSA focus on glenohumeral relationships, such as repairing the subscapularis, increasing humeral component anteversion, and preventing impingement between the humeral polyethylene and the scapular neck. However, IR is a complex shoulder movement involving motion beyond the glenohumeral joint, including scapulothoracic, sternoclavicular, acromioclavicular, and truncal motion.

Studies evaluating shoulder girdle mechanics during abduction and forward elevation after RSA have shown increased dependence on scapulothoracic motion to compensate for less glenohumeral motion. Furthermore, Sulkar et al. performed bi-plane fluoroscopy to compare shoulder kinematics in low and high IR performers after RSA. Patients in the high rotation group had 7° greater scapular upward rotation and used a 15°-30° change in scapular tilt to perform IR in adduction, whereas tilt barely changed (<5°) in most patients in the low group. Interestingly, scapular notching occurred at similar rates in high and low performing cohorts, suggesting that scapular motion can compensate for bony impingement at the glenohumeral joint.

It stands to reason that a prehabilitation program focused on strengthening internal rotators and improving patients' neuromuscular control of the scapula may enable them to adapt more effectively to the altered biomechanics of RSA, and improve their ability to perform ADLs that require IR. Previous studies have demonstrated a moderate correlation between patients' preoperative shoulder strength and range of motion and their postoperative function. However, to date, no studies have attempted to determine whether preoperative improvement in shoulder mobility and strength might confer a durable improvement in shoulder function after RSA, particularly in IR. In the lower extremity, meta-analyses of randomized controlled trials of the total knee arthroplasty literature have found superior knee range of motion and sit-to-stand test performance in patients that underwent a prehabilitation program compared to controls.

The overarching objective is to assess the impact of prehabilitation IR strengthening and mobility on patients undergoing RSA. The specific aim of this study is to determine whether a preoperative rehabilitation program aimed at strengthening shoulder internal rotators and improving scapular mobility can improve patient-reported ability to perform IRADLs postoperatively, as evaluated using the Activities of Daily Living which require Internal Rotation (ADLIR) score.

Hypothesis 1: The investigators hypothesize that patients randomized to the treatment group (IRTx) will have significantly higher ADLIR scores than the control subjects (SOC), postoperatively.

Hypothesis 2: The investigators hypothesize that patients in IRTx group will have greater internal rotation ROM and strength postoperatively as compared to the SOC group.

Data Collection: After informed consent is obtained, all subjects will be randomized 1:1 into treatment (IRTx) or control (COS) cohorts. Randomization will be determined by using a commercial random number generator. Subjects will also have their RSA scheduled approximately 6-8 weeks after enrollment to allow sufficient time for subjects randomized to the IRTx group to complete the preoperative rehabilitation program.

All subjects will attend two in-person sessions at the UF Health Hand and Upper Extremity Rehab Center at the Orthopaedic Sports Medicine Institute for evaluative testing of their shoulder by a trained Physical or Occupational Therapist. The initial visit will occur approximately 6-8 weeks prior to surgery with the second visit occurring 6 weeks later, coinciding with their standard of care pre-operative visit with their surgeon that occurs around 2 weeks prior to surgery.

Shoulder arthroplasty patients undergo routine shoulder range of motion and strength testing during their pre-operative and post-operative clinical visits with their shoulder surgeon and therapist as part of standard of care. For this study, subjects will undergo an additional testing session at the initial visit with their therapist 6 weeks prior to their standard of care pre-operative visit. Range of motion is measured with a standard goniometer. Strength measures are obtained using a hand-held dynamometer (Lafeyette Instruments, Lafayette, IN, USA). These objective measures from both pre-operative visits and visits up to 2 years post-surgery will be collected and used for analysis.

All shoulder arthroplasty patients also complete a self-reported pain, function and general health status questionnaire as part of standard of care both before and at various timepoints after surgery. The Upper Extremity Long Questionnaire used by our clinicians allows the examiner to derive the following scores: Shoulder Pain and Disability Index (SPADI), Simple Shoulder Test (SST-12), American Shoulder and Elbow Surgeons Questionnaire (ASES), UCLA Shoulder Score (UCLA), Short Form Health Survey (SF-12), Constant Shoulder Score and the Shoulder Arthroplasty Smart Score (SAS). These scores up to 2 years post-surgery will be collected for use in this study. Additionally, enrolled subjects will be asked to complete the Activities of Daily Living which require Internal Rotation (ADLIR) questionnaire described by Werthel et al. The investigators believe evaluating patient-reported IR to be a better outcome measure than attempting to objectively measure IR because there exists a known discrepancy between objective IR and patient-reported ability to perform many activities of daily living. This score has been validated for RSA with high internal validity. The ADLIR questionnaire will obtained at both of the subjects' preoperative therapy visits and post-operatively at 12 weeks, 6 months (if applicable), 1 year and 2 years.

Subjects will also have their baseline data collected from their medical record and the shoulder arthroplasty clinical database including demographics, complete medical history including shoulder surgical history and co-morbidities, diagnosis, and radiographic findings. Following surgery the investigators will collect intraoperative findings (e.g., status of the rotator cuff), technical details related to surgery (e.g., use of preoperative planning and surgical navigation, implants characteristics, repair of the subscapularis muscle), length of surgery, surgical complications, post-surgical reoperation/revision, and radiographic outcomes. A complete list of data points is listed on the attached data sheet.

Prehabilitation Protocol:

During the initial therapy visit, subjects randomized to the IRTx cohort will also be instructed by a Physical or Occupational Therapist to perform the exercises described in the attached RSA IR Prehab Exercise Protocol handout, 5-7 times per week for 6 weeks. These exercises are commonly prescribed to patients following shoulder surgery to improve internal range of motion and scapular stabilization. Subjects will be provided with an exercise log to keep track of their progress each week. The research team will inquire about the subjects' progress and exercise logs weekly via a personalized link through REDCaps' text message and email platform, or through phone calls conducted by the research study team. The logs will be collected at the conclusion of the prehabilitation exercise program at the second therapy visit.

Data Analysis:

Data collected for the specific aim and two hypotheses will be analyzed using R Software. First, data will be reviewed for missing entries; in such cases, single imputation using the random forest method (missForest package in R) will be used with patient demographic information, surgical characteristics, and outcome data from all available visits used to inform the model. After missing data has been remedied and continuous measures will be summarized as means and standard deviations. Categorical measures will be summarized as counts and percentages. The SOC and IRTx group demographics and clinical results will be compared for differences with use of Fisher's Exact test and Welch's t-test. Towards our primary outcome, Welch's two-sided t-test will be used to evaluate whether patients who underwent the prehabilitation program achieved more favorable ADLIR scores. Secondary outcomes will be evaluated using the appropriate statistical tests; in most cases, this will consist of Welch's t-test.

Data Management:

Upon enrollment, subjects will be assigned a unique subject research identification number. Once all subject data is collected, PHI will be removed from the data files, and the data will be maintained by using the assigned research subject identification number in preparation for analysis. Dates will also be converted to time frames. A separate key code will be kept until the end of the study.

Data will be maintained in a REDCap database and in an excel database that will be stored on a password-protected encrypted server located in the Department of Orthopaedic Surgery and Sports Medicine and/or Microsoft Teams folder only accessible by study team members. Data analysis will also be stored on this server with only the study team members having access to these files. Paper and pencil questionnaires and exercise logs will be stored in a locking file cabinet. Data will be used only in aggregate and no identifying characteristics of individuals will be published or presented. After the study is completed, the key code will be destroyed, and local data will be stored with other completed research studies in a secured storage room until the appropriate time when the research files may be purged according to university policy.

ELIGIBILITY:
Inclusion Criteria: • Patients aged 40-80

* Undergoing primary RSA for glenohumeral osteoarthritis or rotator cuff arthropathy
* Must be able to read and speak English
* Willing and able to attend a monthly therapy session and perform exercises at home for a minimum of 6 weeks before surgery
* Willing and able to participate in postoperative monitoring for a minimum of 2 years

Exclusion Criteria:

* Patients under the age of 40 and over the age of 80.
* Diagnosis of septic shoulder, fracture, or fracture sequelae, or tumor pathology of the ipsilateral shoulder
* Pre-existing hand, wrist, or elbow pathology that limits elbow flexion or extension, or forearm pronation or supination
* Planned to undergo synchronous procedure of the involved extremity (e.g., synchronous RSA and carpal tunnel release)
* Tendon transfer (e.g., Latissimus dorsi transfer) performed intraoperatively
* Patients without access to phone or email communication for at least 2 years after treatment
* Revision shoulder arthroplasty

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those patients who are indicated for primary reverse total shoulder arthroplasty with one of the attending surgeons on the study team that meet the inclusion/exclusion criteria will be approached by study team members to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living which require Internal Rotation (ADLIR) questionnaire | 6-8 Weeks pre surgery, 2 Weeks pre surgery, and 12 weeks, 6 months, 1 year, 2 years post surgery
  Activities of Daily Living questionnaire with a scale of 9 = worst, 100 = best
  Shoulder Internal Range of Motion Measurements with scoring scale:
  0 = Thigh or less.1 = Hip. 2 = Buttocks, 3 =Sacrum, 4 = L4-L5, 5 = L1-L3, 6 = T12-T8, 7 = T7 or Higher

SECONDARY OUTCOMES:
Shoulder Internal Range of Motion Measurements | 6-8 Weeks pre surgery, 2 Weeks pre surgery, and 12 weeks, 6 months, 1 year, 2 years post surgery
  Higher score the better and equates to better range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Department of Orthopaedics and Rehabilitation, Gainesville, Florida, United States